CLINICAL TRIAL: NCT01549041
Title: A Randomized Comparison of Twice-Daily Versus Once-Daily Asenapine for Schizophrenia
Brief Title: Once-Daily Asenapine for Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00029068
Record Dates: First submitted 2011-10-14; First posted 2012-03-08 (Estimated); Results first posted 2014-05-26 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2013-11

CONDITIONS: Schizophrenia
Keywords: schizophrenia; asenapine; Once daily; twice daily
MeSH Terms: conditions — Schizophrenia | interventions — asenapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- asenapine 10 mg daily in the evening (Experimental): Patients will receive their entire daily dose of asenapine as a single dose in the evening
  Interventions: Drug: Asenapine 10 mg daily in the evening
- asenapine 5 mg twice daily (Active Comparator): Patients will receive asenapine 5 mg daily in the morning and 5 mg daily in the evening
  Interventions: Drug: Asenapine 5 mg twice daily

INTERVENTIONS:
Drug: Asenapine 10 mg daily in the evening — The total daily dose of Asenapine will be given once daily in the evening
  Other Names: Saphris
  Arms: asenapine 10 mg daily in the evening
Drug: Asenapine 5 mg twice daily — Asenapine will be given in two doses, 5 mg in the morning and 5 mg in the evening, daily
  Other Names: Saphris
  Arms: asenapine 5 mg twice daily

SUMMARY:
The investigators propose to explore: 1. the acceptance by patients of once versus twice daily dosing with asenapine, 2. the acceptance by staff of once versus twice daily dosing with asenapine, and 3. the changes in psychopathology associated with these two dosing strategies, in 30 patients with schizophrenia or schizoaffective disorder.

The investigators hypothesize that patient and staff acceptance will be better with once daily dosing and that improvements in psychopathology will be similar across once daily and twice daily dosing

DETAILED DESCRIPTION:
The investigators will randomly assign 30 patients newly admitted to Central Regional Hospital (CRH) for a psychotic exacerbation of schizophrenia or schizo-affective disorder to 14 days of treatment with either asenapine 5 mg BID or asenapine 10 mg QHS.

The investigators will assess patient and staff acceptance on day 14. The investigators will assess staff acceptance on day 14. The investigators will assess changes in psychopathology (Brief Psychiatric Rating Scale) from baseline to day 14.

The investigators propose to achieve the following specific aims:

1. To compare the patient acceptance of once daily versus twice daily asenapine; The investigators hypothesize that patient acceptance will be better for asenapine 10 mg QHS than for asenapine 5 mg BID at day 14
2. To compare the staff (medication nurses) acceptance of once daily versus twice daily asenapine; the investigators hypothesize that staff acceptance will be better for asenapine 10 mg QHS than for asenapine 5 mg BID at day 14
3. To compare the changes in psychopathology with once daily versus twice daily asenapine; the investigators hypothesize that changes in psychopathology from baseline to day 14 will be similar for the two dosing strategies

ELIGIBILITY:
Inclusion Criteria:

* Male or female individuals,
* 18-65 years of age,
* who meet DSM-IV diagnostic criteria for schizophrenia or schizoaffective disorder,
* who are newly admitted to Central Regional Hospital for treatment of an acute psychotic exacerbation,
* who provide signed informed consent to participate, will be included.

Exclusion Criteria:

* Females who are lactating or pregnant,
* individuals with a prior history of poor therapeutic response or sensitivity to asenapine, will be excluded

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Beyer, MD, Principal Investigator — Duke University
Locations (1):
- Central Regional Hospital, Butner, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 30 PATIENTS PARTICIPATED AND WERE RANDOMIZED 12 WERE RANDOMIZED TO ASENAPINE 10 MG QHS 18 WERE RANTOMIZED TO ASENAPINE 5 MG BID
Groups:
- Asenapine 10 mg Daily in the Evening: Patients will receive their entire daily dose of asenapine as a single dose in the evening
  Asenapine 10 mg once daily in the evening: The total daily dose of Asenapine will be given once daily in the evening
Period: Overall Study
Arm/Group | Asenapine 10 mg Daily in the Evening | Asenapine 5 mg Twice Daily
Started | 12 | 18
Completed | 10 | 10
Not Completed | 2 | 8
Not completed — Lack of Efficacy | 2 | 4
Not completed — Adverse Event | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Asenapine 10 mg Daily in the Evening | Asenapine 5 mg Twice Daily | Total
Number analyzed (Participants) | 12 | 18 | 30
Age, Continuous [Mean (Full Range); unit: years]
  age | 41.2 [22 to 61] | 33.1 [20 to 56] | 36.3 [20 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 5 | 8 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 14 | 24
  White | 1 | 4 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 18 | 30

OUTCOME MEASURES:

1. Primary Outcome: Patient Acceptance
Description: A Patient Acceptance Likert Scale (1= Very Acceptable to 7 = Completely Unacceptable, i.e., individual refuses further doses) will be administered to the patient by the Research Nurse on day 14 of treatment.
Time Frame: At day 14
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Asenapine 10 mg Daily in the Evening | Asenapine 5 mg Twice Daily
Number analyzed (Participants) | 12 | 18
units on a scale | 1.7 (0.5) | 3.9 (0.5)

2. Secondary Outcome: Change in Brief Psychiatric Rating Scale (BPRS) Total Score
Description: The BPRS will be completed by the Principle Investigator at baseline and at day 14. The BPRS has 18 items each rated 1-7 with 1 representing the lowest severity of symptoms and 7 representing the highest severity; thus the lowest and highest possible total scores are 18 and 126
Time Frame: From baseline to day 14
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Asenapine 10 mg Daily in the Evening | Asenapine 5 mg Twice Daily
Number analyzed (Participants) | 12 | 18
units on a scale | 16.08 (2.64) | 7.72 (2.21)

ADVERSE EVENTS:
Arm/Group | Asenapine 10 mg Daily in the Evening | Asenapine 5 mg Twice Daily
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/18
Other Adverse Events (participants affected / at risk) | 0/12 | 4/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asenapine 10 mg Daily in the Evening (N=12) | Asenapine 5 mg Twice Daily (N=18)
daytime drowsiness (Nervous system disorders) | 0 (0) | 4 (4) — excessive sedation during the day

LIMITATIONS AND CAVEATS:
Small sample size Open label design

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No